CLINICAL TRIAL: NCT04895995
Title: Initial Assessment of the Feasibility and Efficacy of a Scalable Digital CBT for Generalized Anxiety and Associated Health Behaviors in a Cardiovascular Disease Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6035E
Record Dates: First submitted 2021-05-05; First posted 2021-05-21 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Anxiety Disorders; Cardiovascular Diseases; Anxiety; Health Behavior
MeSH Terms: conditions — Anxiety Disorders; Cardiovascular Diseases; Health Behavior

STUDY DESIGN:
Intervention Model Description: The allocation scheme below refers to Phase 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Cognitive Behavior Therapy (dCBT) for Generalized Anxiety Disorder (Experimental)
  Interventions: Behavioral: Daylight dCBT Application
- Waitlist Control (No Intervention)

INTERVENTIONS:
Behavioral: Daylight dCBT Application — Participants will complete up to four modules of digital intervention delivered in a self-paced format.
  Other Names: Daylight
  Arms: Digital Cognitive Behavior Therapy (dCBT) for Generalized Anxiety Disorder

SUMMARY:
The treatment of generalized anxiety disorder (GAD) in an accessible manner represents an unmet need for those with cardiovascular disease (CVD), given that patients with CVD experience numerous barriers for in-person treatment engagement. The research plan for the proposed pilot project will entail: (1) open study of the acceptability of the digital intervention (N=5), followed by (2) recruitment and randomization of 90 individuals with a history of acute CVD events and clinical levels of GAD symptoms to dCBT or a waitlist (Control) condition, using a 1.5:1 allocation (dCBT:Control).

DETAILED DESCRIPTION:
The treatment of generalized anxiety disorder (GAD) in an accessible manner represents an unmet need for those with cardiovascular disease (CVD), given that patients with CVD experience numerous barriers for in-person treatment engagement. A recent large-scale efficacy trial of digital cognitive behavior therapy (dCBT) for GAD demonstrated significant benefit relative to waitlist control with a large effect size. The research plan for the proposed pilot project will entail: (1) open study of the acceptability of the digital intervention, followed by (2) recruitment and randomization of 90 individuals with a history of acute CVD events and clinical levels of GAD symptoms to dCBT or a waitlist (Control) condition, using a 1.5:1 allocation (dCBT:Control). Assessments will occur at Week 0 (baseline), Week 3, Week 6, and Week 10 (post-treatment).

ELIGIBILITY:
Inclusion Criteria:

* Experienced an acute CVD event (i.e., myocardial infarction, stroke/transient ischemic attack, cardiac arrest, unstable angina, congestive heart failure with hospitalization; exclusion of coronary heart disease, atrial fibrillation, and other arrhythmias)
* Clinical levels of GAD symptoms as operationalized by a score of ≥10 on the GAD-7
* Age 18 or older.
* Individuals must be in the post-acute phase of their CVD; this is operationalized as > 2 months post an acute cardiac event.

Exclusion Criteria:

* Non-English speaker/literate
* No access to a digital device
* Severely vision impaired
* Severe cognitive impairment
* Pending acute surgery or with a life prognosis of fewer than 6 months
* The presence [by self-report] of schizophrenia, psychosis, bipolar disorder, seizure disorder, or current substance use disorder other than nicotine
* Initiation or change of psychotropic medication dosage within the past 4 weeks
* Received CBT for anxiety in last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder Scale (GAD-7) | Week 10 (post-treatment)
  Well validated self-report measure of generalized anxiety disorder symptoms. Scores can range from 0 to 21 with higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Cardiac Anxiety Questionnaire Fear Subscale (CAQ-Fear) | Week 0, Week 6, and Week 10 (post-treatment)
  Well validated 8-item measure of heart-related fear and worry. Scores can range from 0 to 32 with higher scores indicating greater cardiac anxiety.
Smoking History Questionnaire | Week 0, Week 6, and Week 10 (post-treatment)
  Measure of the frequency and amount of recent cigarette use and motivation to quit.
International Physical Activities Questionnaire (IPAQ) | Week 0, Week 6, and Week 10 (post-treatment)
  Well validated self-report measure of how many minutes a day and days a week an individual spends engaged in physical activity.
World Health Organization (WHO) STEPS Instrument - Consumption of Fruit and Vegetables | Week 0, Week 6, and Week 10 (post-treatment)
  Number of servings per day of fruit and vegetables measured by relevant questions on the WHO STEPS Instrument.
Modified Morisky Scale | Week 0, Week 6, and Week 10 (post-treatment)
  This measures will be used to determine medication adherence. Scores can range from 0 to 6 with higher scores indicating greater adherence.
Center for Epidemiological Studies Depression Scale 10 Item Version | Week 0, Week 6, and Week 10 (post-treatment)
  Validated 10-item self-report measure of depression symptoms. Scores can range from 0 to 30 with higher scores indicating greater depression.
Sleep Condition Indicator (SCI-8) | Week 0, Week 6, and Week 10 (post-treatment)
  This 8-item self-report measure is widely used to characterize sleep quality. Scores can range from 0 to 32 with higher scores indicating greater sleep difficulties.
Short Form Health Survey (SF-12) | Week 0, Week 6, and Week 10 (post-treatment)
  This 12-item measure is widely used to evaluate quality of life related to both physical and mental health with cardiac patients. Scores for each subscale range from 0 to 100 with higher scores indicating greater physical and mental health.
Anxiety Sensitivity Inventory (ASI-3) | Week 0, Week 6, and Week 10 (post-treatment)
  This 16-item self-report measures evaluates individuals' tendency to fear and perceive anxiety-related sensations as harmful. Scores can range from 0 to 72 with higher scores indicating greater anxiety sensitivity.
Penn State Worry Questionnaire (PSWQ) | Week 0, Week 6, and Week 10 (post-treatment)
  The PSWQ is the most commonly used self-report measure of worry in research on CBT and dCBT. Scores can range from 16 to 80 with higher scores indicating greater worry.
Shame Inventory-Part 1 (SI-P1) | Week 0, Week 6, and Week 10 (post-treatment)
  This 3-item self-report measures assesses the frequency, intensity, and adverse effects of shame related to physical and mental health. Scores can range from 0 to 12 with higher scores indicating greater shame.
Generalized Anxiety Disorder Scale (GAD-7) | Week 0, Week 3, Week 6
  Well validated self-report measure of generalized anxiety disorder symptoms. Scores can range from 0 to 21 with higher scores indicating greater anxiety.
Resolution of Clinical GAD | Week 10 (post-intervention)
  The proportion of patients no longer meeting GAD-7 clinical severity, operationalized as a score of less than 10 at the 10 week evaluation. Scoring will be the same as described for the GAD-7 above.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parsons EM, Hiserodt M, Otto MW. Initial assessment of the feasibility and efficacy of a scalable digital CBT for generalized anxiety and associated health behaviors in a cardiovascular disease population. Contemp Clin Trials. 2023 Jan;124:107018. doi: 10.1016/j.cct.2022.107018. Epub 2022 Nov 19. PMID 36414206